CLINICAL TRIAL: NCT03249025
Title: Ambulatory Infusion of Lidocaine and Ketamine for Management of Chronic Pain: An Observational Prospective Study
Brief Title: Lidocaine-Ketamine for Management of Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Michael Gofeld, Anesthesiologist, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGD-002-20170705
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Chronic Pain Syndrome
Keywords: lidocaine; ketamine; infusion
MeSH Terms: interventions — Lidocaine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lidocaine-Ketamine Infusion (Experimental): Lidocaine-Ketamine Infusions 1 time per month for 6 months. Pretreatment with Midazolam 1-3 mg IV Push or Subcutaneously and Clonidine 0.1 mg PO prior to infusion.
  Interventions: Drug: Lidocaine; Drug: Ketamine

INTERVENTIONS:
Drug: Lidocaine — Initial dose of 5.0 mg/kg (based on actual weight, up to maximum dose 600 mg) over 45-60 minutes, followed by increases of 0.5 mg/kg each infusion based on tolerability of side effects, to a maximum total dose of 600 mg. The initial and subsequent dose may be increased or decreased by 20% based on patient comorbidities, age and previous experience
Drug: Ketamine — initial dose of 0.25 mg/kg (based on actual weight) over 45-60 minutes (rounded to nearest 5 mg), increased by 10mg each infusion based on tolerability of side effects. The initial and subsequent dose may be increased or decreased by 20% based on patient comorbidities, age and previous experience

SUMMARY:
Chronic pain is defined as 'an unpleasant sensory and emotional experience associated with actual or potential tissues damage, or described in terms of such damage". It is estimated that 1 in 5 Canadians experience chronic pain "Chronic pain is associated with the worst quality of life compared with other chronic diseases such as chronic lung or heart disease". Many of these problems are confined to a specific anatomic structure, and can be diagnosed and treated by injections, physical therapy, surgery, etc. Nonetheless, other individuals experience a more generalized pain. This condition has also resulted I depressed mood, bad relations with other people, sleep disturbances and poor quality of life.

The condition is very difficult to manage, and multiple methods have been recommended. Therapeutic intravenous infusion may be considered as one of these methods. Patients come for infusions of non-opioid medications under medical supervision and in a scheduled fashion. Two most commonly used mediation are lidocaine and ketamine.

Even though it is common to use multiple medications with complementary mechanisms of action to treat pain a combined lidocaine-ketamine infusion has never been studied Therefore, the purpose of this research study is to determine whether mixture of two medications (ketamine and lidocaine) infused intravenously 1 time per month for 6 months results in reduction of pain unpleasantness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Pain duration: > 3 months
* Multifocal and/or non-dermatomal neuropathic pain per Pain Diagram
* Failed medical management with at least 2 neuromodulation agents (e.g., gabapentinoids, antidepressants)
* Neuropathic component (>15 points on S-LANSS)

Exclusion Criteria:

* Non-English speakers
* Refusal to sign informed consent
* Body weight > 100 kg
* Allergies to ketamine and/or lidocaine
* Known contraindications to ketamine use which include poorly controlled systemic illnesses: arterial hypertension, hyperthyroidism, ischemic heart disease, heart failure, psychiatric comorbidity (e.g., history of psychosis, schizophrenia, dissociative state).
* Known contraindication to lidocaine use which include current symptomatic or clinically significant brady- or tachyarrhythmia, systolic blood pressure <90 or >180 mmHg.
* Scheduled interventions targeting neuropathic pain: epidural injections, peripheral nerve blocks, Bier block, radiofrequency of dorsal root ganglia and peripheral nerves, additional lidocaine or ketamine infusions
* Newly added analgesic or neuromodulating medications, or recently performed interventions including lidocaine infusions (in the previous 3 months), or previous lidocaine/ketamine infusion in the previous 360 days. -Acute intoxication or active illegal substance abuse (excluding marijuana)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Unpleasantness Score | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Relative change on "Pain Unpleasantness Score". Moderate clinically important improvement is considered as 30% reduction.

SECONDARY OUTCOMES:
Pain Interference | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Less Pain Interference measured by Short Form Brief Pain Inventory (SF-BPI)
Neuropathic Pain | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Less Neuropathic pain measured by Self-Administered the Leads Assessment of Neuropathic Symptoms and Signs (S-LANSS)
Functional Status | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Improved Functional Status measured by Patient Self-Efficacy Questionnaire (PSEQ)
Emotional Status | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Improved Emotional Status measured by Beck Depression Inventory (BDI), Pain Catastrophizing Scale (PCS)
Cognitive Status | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  No change in Cognitive Status measured by Montreal Cognitive Assessment (MoCA)
Quality of Life | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Improved Quality of Life measured by Global Improvement and Satisfaction Score
Health Care Utilization | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Less Health Care Utilization measured by Self-report of number of physician, clinic visits for other reason, emergency department visit and hospitalizations
Medication Use | Baseline, 1, 2, 3, 4, 5, 6 and 12 Months
  Less Medication Use determined by Type and Dose of medications

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gofeld, MD, FRCPC, Principal Investigator — Michael G. DeGroote Pain Clinic, Hamilton Health Sciences

IPD SHARING:
Plan to Share IPD: No